CLINICAL TRIAL: NCT06309654
Title: Home-Based Circuit Training Attenuates Cardiovascular Risk and Amplifies Functionality and Quality of Life in Overweight/Obese Older Adult Patients With KOA and Type 2 Diabetes: A Randomized Controlled Trial During the COVID-19
Brief Title: Home-Based Circuit Training in Overweight/Obese Older Adult Patients With Knee Osteoarthritis and Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Princess Nourah Bint Abdulrahman University (Other)
Responsible Party: Principal Investigator, Monira Aldhahi, Associate professor, Princess Nourah Bint Abdulrahman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PNU
Record Dates: First submitted 2024-03-01; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Aerobic Exercise; Strength Training; Glycemic Control; Blood Pressure; Oxidative Stress; Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Seventy overweight or obese patients with KOA and T2DM (62.2 ± 6.1 years; 56% female) were randomly assigned to the intervention group (n = 35, HBCT) or the no-exercise control group (n = 35, CON). HBCT performed a progressive protocol (seven exercises; 15-30 repetitions per exercise, 1 min passive rest between exercises; 2-4 rounds per session; 20-60 min total session duration). The knee injury and osteoarthritis symptoms, cardiovascular and metabolic risk factors, cardiorespiratory fitness, and renal function were assessed at baseline and following the 12-week intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- home-based circuit training (HBCT) protocol (Experimental): Participants in the exercise group performed HBCT three times per week on non-consecutive days for 12 weeks.
  Interventions: Behavioral: 12-week home-based circuit training (HBCT)
- Standard of care (CONT) (Sham Comparator): Providing education about the nature of OA, its progression, and strategies for symptom management.
  Empowering individuals with self-management techniques, such as joint protection strategies, activity modification, and lifestyle changes (e.g., weight management, exercise).
  Interventions: Behavioral: Standard of care (CONT)

INTERVENTIONS:
Behavioral: 12-week home-based circuit training (HBCT) — Participants in the exercise group performed HBCT three times per week on non-consecutive days for 12 weeks. The first session was conducted at USM Hospital and participants were instructed how to perform the prescribed exercises in a correct form. In each session, participants performed seven exercises (two aerobic- and five resistance-based) in a circuit fashion, using bodyweight movements and adjustable dumbbells for varied weights, activating all the major muscle groups. In weeks 1-6, participants executed 15 repetitions for 2 rounds with 1 min passive rest between exercises and rounds. In weeks 7-12, participants executed 30 repetitions for 4 rounds with the same rest as prescribed in weeks 1-6. Each round lasted 10-15 min and the total session duration was 20-60 min, aiming to help participants adapt gradually to increasing training volume.
  Arms: home-based circuit training (HBCT) protocol
Behavioral: Standard of care (CONT) — Providing education about the nature of OA, its progression, and strategies for symptom management.
  Empowering individuals with self-management techniques, such as joint protection strategies, activity modification, and lifestyle changes (e.g., weight management, exercise).
  Arms: Standard of care (CONT)

SUMMARY:
Background: Obesity and type 2 diabetes mellitus (T2DM) are considered two of the most prevalent metabolic diseases linked to the onset of knee pain caused by osteoarthritis. Regular exercise has been documented as a principal component of a prevention, management, and treatment strategy for knee osteoarthritis (KOA) patients. However, evidence-based exercise protocols for individuals with comorbidities such as obesity, T2DM, and KOA are scarce. Thus, the present pragmatic randomized controlled trial aimed to investigate the effectiveness of a 12-week home-based circuit training (HBCT) protocol on various indicators related to KOA and cardiometabolic health among overweight/obese older adult patients with KOA and T2DM during the COVID-19 lockdown. Methods: Seventy overweight or obese patients with KOA and T2DM (62.2 ± 6.1 years; 56% female) were randomly assigned to the intervention group (n = 35, HBCT) or the no-exercise control group (n = 35, CON). HBCT performed a progressive protocol (seven exercises; 15-30 repetitions per exercise, 1 min passive rest between exercises; 2-4 rounds per session; 20-60 min total session duration). The knee injury and osteoarthritis symptoms, cardiovascular and metabolic risk factors, cardiorespiratory fitness, and renal function were assessed at baseline and following the 12-week intervention. Results: HBCT significantly improved HBCT improved the vast majority of outcomes related to cardiometabolic health and knee osteoarthritis symptoms compared to CON (p<0.05). No significant differences were detected in total bilirubin, sodium, urea, resting heart rate, or KOOS-sport between HBCT and CON. Conclusion: These findings suggest that an injury-free HBCT program may improve several cardiometabolic health- and KOA-related indices in overweight/obese patients with T2DM and KOA. Such results may encourage clinicians and practitioners to adopt real-world exercise training approaches when prescribing physical exercise to patients characterized by impaired metabolic and musculoskeletal health.

DETAILED DESCRIPTION:
Introduction Despite the beneficial exercise training-induced adaptations, the optimal exercise strategy for populations with obesity, T2DM, and knee osteoarthritis (KOA) presents with some shortcomings in the current literature. More importantly, there are no explicit exercise recommendations in the current KOA guidelines (Kolasinski et al. 2020). Hence, this pragmatic trial was carried out in a home-based setting, aiming to principally investigate the effectiveness of a 12-week home-based circuit training (HBCT) protocol on various outcomes related to knee osteoarthritis symptoms and cardiometabolic health among previously inactive, overweight/obese older adult patients with KOA and T2DM in the real world.

Methods A total of 35 participants were required for this study after considering a dropout rate of 20%. This study involved 69 patients meeting the inclusion criteria as follows: i) age >55 years, ii) diagnosed with KOA with Kellgren-Lawrence criteria grades 2 and 3, indicating moderate KOA, which was based on radiological assessments conducted by a traumatologist, iv) chronic knee pain for more than three months, v) T2DM based on fasting plasma glucose >7.0 mmol·L-1 and glycated hemoglobin (HbA1c) >6.5%, vi) overweight or obesity (BMI ≥25 kg/m2), vii) receiving the standard treatment (all patients were taking diabetes medications), and viii) providing a certificate of a negative COVID-19 diagnostic test (PCR or rapid test). Patients were excluded from the study if during the intervention they demonstrated i) secondary KOA, ii) acute knee pain, iii) changes in medication, supplementation, and/or diet, iv) changes in habitual physical activity, v) intraarticular hyaluronic acid injection treatment within one year, vi) smoking, vii) dementia or any psychiatric diseases, viii) adherence to less than 90% of total prescribed exercise sessions, or ix) they tested positive for COVID-19. After informed written consent, patients were asked not to engage in any other forms of exercise and to maintain their current habitual physical activity levels and eating patterns throughout a 3-month intervention period. Thus, the participants' logbook was reviewed at each visit, aiming to ensure that no changes in nutritional behavior and physical activity patterns occurred. CON followed standard treatment (diabetes medications) without engaging in any structured exercise throughout the intervention.

Study design This is a pragmatic randomized controlled trial study registered at the National Medical Research Register (ID: RSCH ID-21-01180-KGTNMRR ID-21-02367-FUM). The patients were recruited via a poster distributed in the Orthopedics Clinic at USM Hospital. Written informed consent was obtained from all participants before the study. Those willing to participate were then selected and randomly assigned to CON or HBCT. More specifically, patients were divided into two groups performed by an independent statistician using computer-generated random allocation sequences

Assessment procedures All patients were instructed to avoid consuming caffeinated beverages and strenuous exercise 24 hours before the first visit. A total of three visits were performed and all outcomes were assessed through the three visits (baseline, weeks 6 and 12). All measurements were performed at USM Hospital. During the first visit (baseline), assessments were carried out for cardiovascular parameters [e.g., resting heart rate (RHR), systolic (SBP) and diastolic (DBP) blood pressure], BMI, biomarkers [e.g., HbA1c, interleukin 6 (IL-6), and superoxide dismutases (SOD)], rate of perceived exertion (RPE), blood oxygen levels (SpO2), and a 6-minute walk test (6MWT) to assess cardiorespiratory fitness (CRF). KOA symptoms and comorbidity score were also assessed. During the second visit at week 6 (mid-testing), an assessment of cardiovascular parameters and KOA symptoms, RPE, SpO2, and 6MWT took place. During the third visit at week 12 (post-testing), similar assessments to those conducted at baseline were carried out.

ELIGIBILITY:
Inclusion Criteria:

* age >55 years
* diagnosed with KOA with Kellgren-Lawrence criteria grades 2 and 3, indicating moderate KOA, which was based on radiological assessments conducted by a traumatologist
* chronic knee pain for more than three months
* T2DM based on fasting plasma glucose >7.0 mmol·L-1 and glycated hemoglobin (HbA1c) >6.5%,
* overweight or obesity (BMI ≥25 kg/m2)
* providing a certificate of a negative COVID-19 diagnostic test (PCR or rapid test).

Exclusion Criteria:

* secondary KOA
* acute knee pain,
* changes in medication, supplementation, and/or diet
* changes in habitual physical activity
* smoking
* dementia or any psychiatric diseases
* adherence to less than 90% of total prescribed exercise sessions
* tested positive for COVID-19

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Blood pressure | end of 12 week
  systolic (SBP) and diastolic (DBP) blood pressure
The A1C test | end of 12 week
blood oxygen levels | end of 12 week
  oxygen level was quantify using SpO2
cardiorespiratory fitness | end of 12 week
  a 6-minute walk test (6MWT)
interleukin 6 (IL-6) | end of 12 week
  an interleukin that acts as both a pro-inflammatory cytokine and an anti-inflammatory myokine will be measured using Human ELISA Kit #P05231 and # P00441, respectively
Superoxide dismutases (SOD) | end of 12 week
  enzyme that alternately catalyzes the dismutation (or partitioning) of the superoxide will be measured using g Plasma IL-6 and SOD levels

CONTACTS AND LOCATIONS:
Overall Officials: Sameer Al-Mhanna, Phd, Study Director — Department of physiology, School of Medical Sciences, Universiti Sains Malaysia, Kubang Kerian 16150, Kelantan, Malaysia
Locations (1):
- Princess Nourah bint Abdulrahman University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No